CLINICAL TRIAL: NCT06143319
Title: The Chronic Pain Brain: Structural White and Gray Matter Correlates of Impaired Muscle Control and Deficient Pain Processing
Brief Title: Structural White and Gray Matter Correlates of Impaired Muscle Control and Deficient Pain Processing
Acronym: B~Maps
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: B670201422908 - EC/2014/1245
Record Dates: First submitted 2022-11-18; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain; Low Back Pain, Recurrent; Low Back Pain, Chronic; Healthy Volunteers; Fibromyalgia
Keywords: low back pain; motor control; central sensitization; brain structure; brain function; central pain processing; fibromyalgia
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Recurrent low back pain: 20 non-specific recurrent LBP patients, both experiencing a period of pain remission or a pain flare at the moment of testing, will be included in the current study.
- Chronic low back pain: 20 participants experiencing non-specific chronic LBP will be included in the current study.
- Healthy volunteers: 20 healthy participants, matched for age and Body Mass Index (BMI) with the participants experiencing chronic/recurrent low back pain or fibromyalgia will be included in the current study.
- Fibromyalgia: 20 participants diagnosed with fibromyalgia will be included in the current study

SUMMARY:
Although the cause of persistent non-specific low back pain (LBP) remains unknown, structural and functional alterations of the brain, alterations in the lumbar muscles and dysfunction of the central nervous system have been proposed as underlying mechanisms. In this case-control study, 1) brain structure/function, 2) lumbar muscle function and 3) central pain processing are compared across four groups: 1) healthy participants, 2) recurrent LBP (both during pain flare and during pain remission), 3) chronic LBP and 4) fibromyalgia. According to previous research, healthy participants and fibromyalgia patients are two extremes of a "musculoskeletal pain continuum". Healthy participants representing one extreme of the continuum with no pain and fibromyalgia representing the other extreme of the continuum with chronic widespread pain. It is thought that different LBP populations (i.e. (sub)acute, recurrent, chronic LBP) float between the aforementioned extremes. Past studies already highlighted the need for studies comparing the pathophysiological mechanisms for different pain syndromes to identify common underlying mechanisms across pain syndromes. For this reason, the goal of the current study is to compare alterations in brain structure/function, alterations in lumbar muscle function and alterations in central pain processing across the aforementioned "musculoskeletal pain continuum". It is hypothesized that longer duration of pain (recurrent vs chronic) and the extensiveness of the pain (one location vs widespread pain) are associated with more pronounced alterations in 1) brain structure/function, 2) lumbar muscle function and 3) central pain processing.

DETAILED DESCRIPTION:
Introduction: Chronic pain is one of the most disabling symptoms in several medical conditions, including LBP and fibromyalgia. A crucial factor for the persistence of recurrent/chronic pain are alterations in lumbar muscle structure and function in patients experiencing recurrent/chronic LBP. Previous studies revealed that these alterations in lumbar muscle structure and function do not resolve when patients with recurrent LBP experience a pain-free episode. According to other recent studies, dysfunction of the central nervous system is another crucial factor to the maintenance of chronic pain. The aforementioned alterations in lumbar muscle structure and function could constitute constant nociceptive input leading to the development of central sensitization (i.e. heightened sensitivity or hyperexcitability of central nervous system). Although it is plausible that central sensitization and disturbed pain processing do exist in patients experiencing chronic LBP, previous studies investigating these mechanisms are scant and results are inconsistent. These inconsistent results might be explained by the fact that previous studies used mixed back pain populations (i.e. different types of back pain are included in one study). In contrast to the inconsistent evidence for the presence of central sensitization in chronic LBP, previous studies in fibromyalgia populations have shown convincing evidence for central sensitization and disturbed pain processing in fibromyalgia. It could be possible that the long-term presence of pain and nociceptive input not only influence pain processing, but also motor control. To support this hypothesis, past studies have revealed altered organization of brain areas involved in trunk and lumbar motor control in patients experiencing recurrent LBP. In addition to alterations in brain function, changes in brain structure are also probable in patients experiencing persistent pain and nociceptive input. Previous studies in fibromyalgia already confirmed the presence of structural brain alterations. To date, only two studies investigated the presence of structural brain alterations in gray matter in patients experiencing LBP and the results are contradicting. Whether structural brain alterations in white matter exist in patients experiencing LBP has not yet explored in previous studies. Past studies in fibromyalgia do confirm that white matter structural changes exist. It is still unclear which specific properties of white matter change in patients with fibromyalgia, because more advanced imaging techniques are necessary to answer this question. In our current study we want to elaborate on the aforementioned results obtained in fibromyalgia patients to investigate whether the same alterations in central mechanisms (i.e. altered pain processing and alterations in brain structure/function) occur in patients experiencing recurrent/chronic LBP. Past studies already highlighted the need for studies comparing similarities and differences in the pathophysiological mechanisms for different pain syndromes to identify similarities in underlying mechanisms across different pain syndromes (e.g. fibromyalgia and LBP). For this reason, the current study will include both patients with fibromyalgia and patients experiencing recurrent/chronic LBP to allow for comparison of the pathophysiological mechanisms.

This case-control study has multiple goals: 1) investigate whether central sensitization and disturbed central pain processing are present in patients experiencing recurrent and chronic LBP. 2) investigate whether structural alterations in gray and white matter exist in patients experiencing recurrent and chronic LBP. 3) investigate whether alterations in white matter microstructure exist in patients experiencing recurrent and chronic LBP and if these alterations are comparable to alterations in white matter structure in fibromyalgia reported in previous studies. 4) investigate whether there is an association between alterations in brain structure/functional connectivity and the degree of disturbances in pain processing. 5) investigate whether there is an association between alterations in brain structure/functional connectivity and lumbar muscle dysfunction. 6) investigate to what extent the duration of pain (i.e. (sub)acute, recurrent, chronic) and the extensiveness of pain (i.e. one location vs widespread pain) influences lumbar motor control, pain processing and brain structure/function.

Method: In this case-control study, 80 female participants will be divided over 4 groups: 1) healthy participants (N=20), 2) recurrent non-specific LBP patients, both during pain remission and during pain flare pain (N = 20), 3) chronic non-specific LBP (N = 20) and 4) fibromyalgia patients (N = 20). The test protocol consists of three parts: 1) participants complete a series of questionnaires measuring several clinical characteristics, including: sociodemographic variables, pain intensity, functional disability, central sensitization and psychosocial factors (i.e. coping, catastrophizing, kinesiophobia, hypervigilance and anxiety/depression). 2) magnetic resonance imaging (MRI) will be used to measure brain structure. Functional MRI (fMRI) and diffusion tensor imaging (DTI) will be used to measure brain function (i.e. resting state and functional connectivity respectively). 3) a series of clinical tests will be performed to measure lumbar muscle function and central pain processing. Lumbar muscle function will be evaluated by using surface electromyography (EMG) for testing anticipatory postural adjustments (APA) in a rapid arm movement (RAM) task and compensatory postural adjustments (CPA) in a quick force release test (QFRT). Central pain processing will be assessed by using 1) pressure algometry for determining pain pressure thresholds (PPT), 2) measuring PPT after a conditioned pain modulation paradigm (CPM) and 3) by determining the nociceptive flexion reflex (NFR) threshold by using repetitive transcutaneous electrical nerve stimulation (TENS) of the n. suralis.

ELIGIBILITY:
Inclusion Criteria:

1. Dutch speaking female participants (age between 18 and 45 years).
2. Non-specific recurrent LBP patients experiencing a period of remission at the moment of testing. Patients have to meet the criteria for recurrent LBP (in remission) as described by De Vet et al. (2002) and D'Hooge et al. (2013).
3. Non-specific recurrent LBP patients experiencing a pain flare at the moment of testing. Patients have to meet the criteria for recurrent LBP (during pain flare) as described by De Vet et al. (2002) and D'Hooge et al. (2013).
4. Participants experiencing non-specific chronic LBP (meeting the International Association for the Study of Pain [IASP] criteria)
5. Participants diagnosed with fibromyalgia according to the American College of Rheumatology (ACR) criteria (2010)
6. Healthy volunteers with no history of serious respiratory, orthopedic, neurologic or circulatory conditions. No history of low back pain (i.e. low back pain in this case is defined as a period of symptoms lasting a minimum of 2 consecutive days and for which a paramedic is consulted). Participants with a history of spinal surgery, spinal trauma or spinal deformities are also excluded. Healthy participants will be matched for age and BMI with included participants experiencing chronic/recurrent LBP or fibromyalgia.

Exclusion Criteria:

1. Pregnancy or breastfeeding in the past year
2. Contraindications for MRI (e.g. electrical/mechanical implants or electrodes in de body, eye/skin injury by metal fragments in the past, etc)
3. BMI lower than 18 or higher than 30
4. Participant performed specific trunk muscle training in the past year.
5. Participating in sports at a professional level

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants are women, recruited through advertisement in hospitals, patient groups and organizations, flyers, social media etc.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Brain structure and function | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  The scanning session will comprise of (1) whole-brain T1-weighted structural MRI, (2) whole-brain DTI and (3) whole-brain resting-state functional MRI (rs-fMRI).
Pressure pain thresholds | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  Pressure algometry for determining the PPT with a digital algometer bilaterally at three body locations, namely on the forearm (on the muscle belly of the extensor carpi radialis muscle), the erector spinae (5cm lateral to the processus spinosus of vertebra L3), and the calf (at the upper third of the distance between the knee crease and the distal border of the calcaneus)
Conditioned pain modulation | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  A CPM paradigm during which the PPT (= test stimulus) is repeated during and after immersion of the non-dominant hand in a warm water bath (= conditioned stimulus) of 45.5°C for six minutes.
Nociceptive flexion reflex thresholds | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  Repetitive TENS of the sural nerve of the dominant leg to determine the NFR threshold and temporal summation of the NFR threshold. A bar stimulating electrode will be connected to a constant current stimulator. Elicitation of the NFR will be evaluated by measuring the involuntary contraction of the ipsilateral biceps femoris.
Lumbar muscle function | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  Lumbar muscle function will be measured by using surface EMG for testing APAs in a RAM test and CPAs in a QFRT.

SECONDARY OUTCOMES:
Pain intensity | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  Pain intensity was measured with two visual analogue scales (0 - 100) for average pain and worst pain. The anchors are 'no pain' and 'unbearable pain' respectively. No grid lines are shown on the scale.
Functional disability | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  To measure functional disability the Dutch version (Beurskens, De Vet et al. 1995) of the Roland and Morris Disability Questionnaire (RMDQ) (Roland and Morris 1983) was used. The RMDQ consists of 24 items, with dichotomous answers: 'Yes' (coded = 1) or 'No' (coded = 0). Scores range from 0-24. Higher scores indicate higher disability.
Coping | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  Coping was measured by using the Dutch version of the Pain Coping Inventory (PCI) (Kraaimaat, Bakker et al. 1997). The PCI consists of 33 questions divided over six subscales: pain transformation, distraction, reducing demands, retreating, worrying and resting (Kraaimaat and Evers 2003). Participants have to rate on 4-point Likert scales to what extend they perform the described behaviors in the statements (e.g. "I take a bath or shower"). Based on the scores of the 33 items, 2 higher order scores are derived for active coping (i.e. transformation, reducing demands, distraction) and passive coping (i.e. retreating, worrying and resting).
Kinesiophobia | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  To measure pain related fear, the Dutch version of the Tampa Scale for Kinesiophobia (TSK) was used (Vlaeyen, Kole-Snijders et al. 1995). The TSK is used to measure the extend of pain-related fear and the influence on activity level in LBP populations. The questionnaire consists of 17 items, with higher scores indicating a higher degree of kinesiophobia. Items are scored on 4-point Likert scales and participants have to rate to what degree they agree/disagree to the statements (e.g. "I'm afraid that I might injure myself if I exercise").
Catastrophizing | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  To measure pain catastrophizing the Dutch version (Crombez 1996) of the Pain Catastrophizing Scale (PCS) was used. The PCS consist of 13 items about past painful experiences. Participants were requested to indicate to what degree they experience certain thoughts or feelings when experiencing pain on a 5-point Likert scale (e.g.: "I worry all the time about whether the pain will end"). The total score ranges from 0-52, with higher scores indicating more pain catastrophizing.
Depression and anxiety | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  To measure symptoms of depression and anxiety, the Dutch version of the Hospital Anxiety and Depression Scale (HADS) was used (Zigmond and Snaith, 1983). The HADS consists of two subscales with 7 items. Scores on both subscales ranges from 0 - 20, with higher scores indicating more anxiety and/or depression. Participants have to indicate on a 4-point Likert scale if they have experienced the emotions described in each statement during the last week (e.g. "I feel restless as I have to be on the move").
Central sensitization | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  The Dutch version of the Central Sensitization Index (CSI) was used to measure for symptoms and clinical features related to central sensitization (i.e. hyperexcitability of the central nervous system) (Kregel, Vuijk et al. 2016). The CSI consists of two parts. The first part measures to what extend somatic and emotional symptoms related to central sensitization are present (e.g. "I get tired very easily when I am physically active") and the second part measures whether participants had earlier diagnosis which are frequently observed in central sensitization of the central nervous system (e.g. fibromyalgia, chronic fatigue syndrome, etc).
Attention to pain | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  To measure attention to pain, the Dutch version of the Pain Vigilance and Awareness Questionnaire (PVAQ) was used (Roelofs, Peters et al. 2003). The PVAQ consists of 16 items with two subscales: 'attention to pain' and 'attention to changes in pain'. Participants have to rate on a 6-point Likert scale to what extend they react in a certain way to pain as described in the statements (e.g. "I am quick to notice changes in pain intensity").
Physical activity | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  The Dutch version of the International Physical Activity Questionnaire (IPAQ) was used to obtain a self-reported estimate of physical activity in the last seven days (Craig, Marshall et al. 2003). The IPAQ consists of 31 items about physical activity divided over 5 areas: job-related, transportation, housework (i.e. house maintenance, caring for family), recreation/sport/leisure and time spent sitting. The overall score places participants in one of three categories: 1) low/inactive, 2) moderately active and 3) highly active.
General health status | The entirety of the protocol for each patient is administered in a single day, spanning approximately 4 to 5 hours.
  To measure general health status and health-related quality of life the Short Form Health Survey-36 items (SF-36) was used (Van der Zee and Sanderman 1993, Aaronson, Muller et al. 1998). The SF-36 measures several domains of health-related areas: physical functioning, physical role limitations, bodily pain, general health perception, energy/vitality, social functioning, emotional role limitations and mental health. Scores range from 0 - 100, higher scores indicating higher subjective health status.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Oosterwijck, Prof, Principal Investigator — Ghent University, Pain in Motion; Lieven Danneels, Prof, Principal Investigator — University Ghent
Locations (1):
- Ghent University, vakgroep revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodges PW, Moseley GL. Pain and motor control of the lumbopelvic region: effect and possible mechanisms. J Electromyogr Kinesiol. 2003 Aug;13(4):361-70. doi: 10.1016/s1050-6411(03)00042-7. PMID 12832166
- [Background] Danneels LA, Coorevits PL, Cools AM, Vanderstraeten GG, Cambier DC, Witvrouw EE, De CH. Differences in electromyographic activity in the multifidus muscle and the iliocostalis lumborum between healthy subjects and patients with sub-acute and chronic low back pain. Eur Spine J. 2002 Feb;11(1):13-9. doi: 10.1007/s005860100314. PMID 11931058
- [Background] Danneels LA, Vanderstraeten GG, Cambier DC, Witvrouw EE, De Cuyper HJ. CT imaging of trunk muscles in chronic low back pain patients and healthy control subjects. Eur Spine J. 2000 Aug;9(4):266-72. doi: 10.1007/s005860000190. PMID 11261613
- [Background] D'hooge R, Cagnie B, Crombez G, Vanderstraeten G, Dolphens M, Danneels L. Increased intramuscular fatty infiltration without differences in lumbar muscle cross-sectional area during remission of unilateral recurrent low back pain. Man Ther. 2012 Dec;17(6):584-8. doi: 10.1016/j.math.2012.06.007. Epub 2012 Jul 10. PMID 22784801
- [Background] D'hooge R, Cagnie B, Crombez G, Vanderstraeten G, Achten E, Danneels L. Lumbar muscle dysfunction during remission of unilateral recurrent nonspecific low-back pain: evaluation with muscle functional MRI. Clin J Pain. 2013 Mar;29(3):187-94. doi: 10.1097/AJP.0b013e31824ed170. PMID 23369927
- [Background] D'hooge R, Hodges P, Tsao H, Hall L, Macdonald D, Danneels L. Altered trunk muscle coordination during rapid trunk flexion in people in remission of recurrent low back pain. J Electromyogr Kinesiol. 2013 Feb;23(1):173-81. doi: 10.1016/j.jelekin.2012.09.003. Epub 2012 Oct 15. PMID 23079004
- [Background] Nijs J, Daenen L, Cras P, Struyf F, Roussel N, Oostendorp RA. Nociception affects motor output: a review on sensory-motor interaction with focus on clinical implications. Clin J Pain. 2012 Feb;28(2):175-81. doi: 10.1097/AJP.0b013e318225daf3. PMID 21712714
- [Background] Roussel NA, Nijs J, Meeus M, Mylius V, Fayt C, Oostendorp R. Central sensitization and altered central pain processing in chronic low back pain: fact or myth? Clin J Pain. 2013 Jul;29(7):625-38. doi: 10.1097/AJP.0b013e31826f9a71. PMID 23739534
- [Background] Meeus M, Nijs J. Central sensitization: a biopsychosocial explanation for chronic widespread pain in patients with fibromyalgia and chronic fatigue syndrome. Clin Rheumatol. 2007 Apr;26(4):465-73. doi: 10.1007/s10067-006-0433-9. Epub 2006 Nov 18. PMID 17115100
- [Background] Tsao H, Danneels LA, Hodges PW. ISSLS prize winner: Smudging the motor brain in young adults with recurrent low back pain. Spine (Phila Pa 1976). 2011 Oct 1;36(21):1721-7. doi: 10.1097/BRS.0b013e31821c4267. PMID 21508892
- [Background] Apkarian AV, Sosa Y, Sonty S, Levy RM, Harden RN, Parrish TB, Gitelman DR. Chronic back pain is associated with decreased prefrontal and thalamic gray matter density. J Neurosci. 2004 Nov 17;24(46):10410-5. doi: 10.1523/JNEUROSCI.2541-04.2004. PMID 15548656
- [Background] Schmidt-Wilcke T, Leinisch E, Ganssbauer S, Draganski B, Bogdahn U, Altmeppen J, May A. Affective components and intensity of pain correlate with structural differences in gray matter in chronic back pain patients. Pain. 2006 Nov;125(1-2):89-97. doi: 10.1016/j.pain.2006.05.004. Epub 2006 Jun 5. PMID 16750298
- [Background] Fayed N, Garcia-Campayo J, Magallon R, Andres-Bergareche H, Luciano JV, Andres E, Beltran J. Localized 1H-NMR spectroscopy in patients with fibromyalgia: a controlled study of changes in cerebral glutamate/glutamine, inositol, choline, and N-acetylaspartate. Arthritis Res Ther. 2010;12(4):R134. doi: 10.1186/ar3072. Epub 2010 Jul 7. PMID 20609227
- [Background] Kang DH, Son JH, Kim YC. Neuroimaging studies of chronic pain. Korean J Pain. 2010 Sep;23(3):159-65. doi: 10.3344/kjp.2010.23.3.159. Epub 2010 Aug 26. PMID 20830260
- [Background] Lutz J, Jager L, de Quervain D, Krauseneck T, Padberg F, Wichnalek M, Beyer A, Stahl R, Zirngibl B, Morhard D, Reiser M, Schelling G. White and gray matter abnormalities in the brain of patients with fibromyalgia: a diffusion-tensor and volumetric imaging study. Arthritis Rheum. 2008 Dec;58(12):3960-9. doi: 10.1002/art.24070. PMID 19035484
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] de Vet HC, Heymans MW, Dunn KM, Pope DP, van der Beek AJ, Macfarlane GJ, Bouter LM, Croft PR. Episodes of low back pain: a proposal for uniform definitions to be used in research. Spine (Phila Pa 1976). 2002 Nov 1;27(21):2409-16. doi: 10.1097/01.BRS.0000030307.34002.BE. PMID 12438991
- [Background] Neziri AY, Curatolo M, Limacher A, Nuesch E, Radanov B, Andersen OK, Arendt-Nielsen L, Juni P. Ranking of parameters of pain hypersensitivity according to their discriminative ability in chronic low back pain. Pain. 2012 Oct;153(10):2083-2091. doi: 10.1016/j.pain.2012.06.025. Epub 2012 Jul 28. PMID 22846347
- [Background] Silfies SP, Mehta R, Smith SS, Karduna AR. Differences in feedforward trunk muscle activity in subgroups of patients with mechanical low back pain. Arch Phys Med Rehabil. 2009 Jul;90(7):1159-69. doi: 10.1016/j.apmr.2008.10.033. Epub 2009 Jun 5. PMID 19501348
- [Background] Nijs J, Inghelbrecht E, Daenen L, Hachimi-Idrissi S, Hens L, Willems B, Roussel N, Cras P, Wouters K, Bernheim J. Recruitment bias in chronic pain research: whiplash as a model. Clin Rheumatol. 2011 Nov;30(11):1481-9. doi: 10.1007/s10067-011-1829-8. Epub 2011 Aug 19. PMID 21853277
- [Background] Wacholder S, Silverman DT, McLaughlin JK, Mandel JS. Selection of controls in case-control studies. III. Design options. Am J Epidemiol. 1992 May 1;135(9):1042-50. doi: 10.1093/oxfordjournals.aje.a116398. PMID 1595690
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Lefever I, Huybrechts L, Lambrecht L, Paul L. Pain inhibition and postexertional malaise in myalgic encephalomyelitis/chronic fatigue syndrome: an experimental study. J Intern Med. 2010 Sep;268(3):265-78. doi: 10.1111/j.1365-2796.2010.02228.x. Epub 2010 Mar 3. PMID 20412374
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Van Loo M, Paul L. Lack of endogenous pain inhibition during exercise in people with chronic whiplash associated disorders: an experimental study. J Pain. 2012 Mar;13(3):242-54. doi: 10.1016/j.jpain.2011.11.006. Epub 2012 Jan 24. PMID 22277322
- [Background] Aaronson NK, Muller M, Cohen PD, Essink-Bot ML, Fekkes M, Sanderman R, Sprangers MA, te Velde A, Verrips E. Translation, validation, and norming of the Dutch language version of the SF-36 Health Survey in community and chronic disease populations. J Clin Epidemiol. 1998 Nov;51(11):1055-68. doi: 10.1016/s0895-4356(98)00097-3. PMID 9817123
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Kraaimaat FW, Evers AW. Pain-coping strategies in chronic pain patients: psychometric characteristics of the pain-coping inventory (PCI). Int J Behav Med. 2003;10(4):343-63. doi: 10.1207/s15327558ijbm1004_5. PMID 14734263
- [Background] Beurskens AJ, de Vet HC, Koke AJ, van der Heijden GJ, Knipschild PG. Measuring the functional status of patients with low back pain. Assessment of the quality of four disease-specific questionnaires. Spine (Phila Pa 1976). 1995 May 1;20(9):1017-28. doi: 10.1097/00007632-199505000-00008. PMID 7631231
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Vlaeyen JWS, Kole-Snijders AMJ, Boeren RGB, van Eek H. Fear of movement/(re)injury in chronic low back pain and its relation to behavioral performance. Pain. 1995 Sep;62(3):363-372. doi: 10.1016/0304-3959(94)00279-N. PMID 8657437
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Kregel J, Vuijk PJ, Descheemaeker F, Keizer D, van der Noord R, Nijs J, Cagnie B, Meeus M, van Wilgen P. The Dutch Central Sensitization Inventory (CSI): Factor Analysis, Discriminative Power, and Test-Retest Reliability. Clin J Pain. 2016 Jul;32(7):624-30. doi: 10.1097/AJP.0000000000000306. PMID 26418360
- [Background] Roelofs J, Peters ML, McCracken L, Vlaeyen JWS. The pain vigilance and awareness questionnaire (PVAQ): further psychometric evaluation in fibromyalgia and other chronic pain syndromes. Pain. 2003 Feb;101(3):299-306. doi: 10.1016/S0304-3959(02)00338-X. PMID 12583873
- See also: Goubert, D. (2017). Peripheral back muscle dysfunctions and central pain mechanisms : an innovative perspective on differences between recurrent and chronic pain. Ghent University. Faculty of Medicine and Health Sciences, Ghent, Belgium. — http://hdl.handle.net/1854/LU-8520794
- See also: Van der Zee, K. and R. Sanderman (1993). "RAND-36." Groningen: Northern Centre for Health Care Research, University of Groningen, the Netherlands 28(6). — https://www.praktijktransire.nl/wp-content/uploads/2022/04/Rand-36-vanaf-pagina-24.pdf
- See also: Kraaimaat, F., A. Bakker and A. Evers (1997). "Pijncoping-strategieën bij chronische pijnpatiënten: De ontwikkeling van de Pijn-Coping-Inventarisatielijst (PCI)." — https://repository.ubn.ru.nl/bitstream/handle/2066/24661/24661.PDF?sequence=1
- See also: Crombez, G. (1996). "De Pain Catastrophizing scale (PCS)." — https://bsw.ugent.be/VVGP/fichePCS.pdf